CLINICAL TRIAL: NCT03307824
Title: A Multicenter Randomized Study on Operative Time When Using IFABOND™ Synthetic Glue in Laparoscopic Sacrocolpopexy
Brief Title: Operative Time During the Use of the Synthetic Glue IFABONDTM in Laparoscopic Sacrocolpopexy
Acronym: Procolle 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0647; 2017-A01405-48 (Other: ID-RCB)
Record Dates: First submitted 2017-10-03; First posted 2017-10-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Prolapse
Keywords: Laparoscopic Surgery; synthetic glue IFABONDTM; time of surgery
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IfabondTM (Experimental): Use of the synthetic glue IfabondTM
  Interventions: Device: Synthetic glue IfabondTM
- sutures (Active Comparator): Glue-Free Suture Technique
  Interventions: Procedure: Glue-Free Suture Technique

INTERVENTIONS:
Device: Synthetic glue IfabondTM — Use of the synthetic glue IfabondTM
  Arms: IfabondTM
Procedure: Glue-Free Suture Technique — Suture Technique
  Arms: sutures

SUMMARY:
Laparoscopic sacrocolpopexy has now become the gold standard technique for correction of anterior and apical prolapse. In order to provide an alternative to stapling system and sutures involving vaginal erosion and shrinkage phenomena, there is a technique to fix material meshes by the use of a liquid, tissue, synthetic adhesive and sterile. The investigator hypothesizes that the use of IFABOND ™ adhesive in laparoscopic sacrocolpopexy significantly reduces the time of surgery compared to the classic suture technique. The prospective, randomized, multicenter study therefore aims to compare the time of surgery when using the IFABOND™ synthetic adhesive and the technique by sutures to fix material meshes in laparoscopic sacrocolpopexy.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18 years or more
* Stage III or IV medial and/or anterior genital prolapse on the Pelvic Organ Prolapse Quantification (POP-Q) classification (hysterocele and/or cystocele) requiring surgical correction
* Patient requesting surgery for the trouble caused by the prolapse

Exclusion Criteria:

* Prolapse of POP-Q stage <III or without functional impact
* Unacceptable postoperative risk disclosed on interview: coagulation disorder, immune disorder, evolutive disease, etc.
* Impaired lower-limb range of motion preventing positioning for surgery
* Pregnancy or intended pregnancy during study period
* Evolutive or latent infection or signs of tissue necrosis on clinical examination
* Non-controlled diabetes (glycated haemoglobin >8%)
* Treatment impacting immune response (immunomodulators), ongoing or within previous month
* History of pelvic region radiation therapy, at any time
* History of pelvic cancer
* Non-controlled evolutive spinal pathology
* Known hypersensitivity to one of the implant components (polypropylene)
* Cyanoacrylate hypersensitivity
* Formaldehyde hypersensitivity
* Inability to understand information provided
* No national health insurance cover; prisoner, or ward of court

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
duration of surgery | Day 0
  time of surgery in minutes (measured by chronometers)

SECONDARY OUTCOMES:
Percentage prolapse correction failure | at 1 months post-surgery
  A correction failure correspond to a patient with stage ≥ II prolapse on the POP-Q classification
Percentage prolapse correction failure | at 12 months post-surgery
  A correction failure correspond to a patient with stage ≥ II prolapse on the POP-Q classification
Percentage prolapse correction failure | at 24 months post-surgery
  A correction failure correspond to a patient with stage ≥ II prolapse on the POP-Q classification
complications | at day 0
complications | at 1 months post-surgery
complications | at 12 months post-surgery
complications | at 24 months post-surgery
pain | at day 0
  assessed by visual analog scale (VAS)
pain | at 1 months post-surgery
  assessed by visual analog scale (VAS)
pain | at 12 months post-surgery
  assessed by visual analog scale (VAS)
pain | at 24 months post-surgery
  assessed by visual analog scale (VAS)
quality of life | at 1 months post-surgery
  assessed by the questionnaires Short Form Health Survey-12 (SF-12)
quality of life | at 1 months post-surgery
  assessed by the questionnaires Pelvic Floor Distress Inventory -20 (PFDI-20)
quality of life | at 1 months post-surgery
  assessed by the questionnaires Pelvic Floor Impact Questionnaire-7 (PFIQ-7)
quality of life | at 1 months post-surgery
  assessed by the questionnaires Patient Global Impression of Improvement (PGI-I)
quality of life | at 12 months post-surgery
  assessed by the questionnaires SF-12
quality of life | at 12 months post-surgery
  assessed by the questionnaires PFDI-20
quality of life | at 12 months post-surgery
  assessed by the questionnaires PFIQ-7
quality of life | at 12 months post-surgery
  assessed by the questionnaires PGI-I
quality of life | at 24 months post-surgery
  assessed by the questionnaires SF-12
quality of life | at 24 months post-surgery
  assessed by the questionnaires PFDI-20
quality of life | at 24 months post-surgery
  assessed by the questionnaires PFIQ-7
quality of life | at 24 months post-surgery
  assessed by the questionnaires PGI-I
sexuality score | at 1 months post-surgery
  assessed by the questionnaire french version of Pelvic Organ Prolapse/Incontinence Sexual Questionnaire (PISQ-12)
sexuality score | at 12 months post-surgery
  assessed by the questionnaire PISQ-12
sexuality score | at 24 months post-surgery
  assessed by the questionnaire PISQ-12
percentage of dyspareunia | at 1 months post-surgery
percentage of dyspareunia | at 12 months post-surgery
percentage of dyspareunia | at 24 months post-surgery
percentage of urinary incontinence | at 1 months post-surgery
percentage of urinary incontinence | at 12 months post-surgery
percentage of urinary incontinence | at 24 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Géry LAMBLIN, MD, Principal Investigator — Gynaecology Department, Hôpital Femme Mère Enfant, HCL
Locations (1):
- Gynaecology Department, Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided